CLINICAL TRIAL: NCT03949387
Title: Functional Electrical Stimulation Cycling for Managing Mobility Disability in People with Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: The Ottawa Hospital (Other); Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Lara Pilutti, Associate Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHSN-REB 20180731-01H
Record Dates: First submitted 2019-05-06; First posted 2019-05-14 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: exercise; multiple sclerosis; mobility
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will use a two-arm, parallel group, single-blinded placebo-controlled RCT design that examines the efficacy and lasting effects of 24-weeks of FES cycling exercise compared to passive leg cycling in persons with MS with mobility impairment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be collected objectively by researchers who are blinded to treatment allocation. Researchers who are involved with delivery of the intervention will be aware of treatment allocation, but will not be involved with data collection, entry or analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FES Cycling Exercise (Experimental): FES cycling will involve systematic, transcutaneous electrical stimulation of the leg muscles to produce leg-cycling movement. The intensity and duration of training will be prescribed based on guidelines for aerobic exercise training for persons with MS and from the American College of Sports Medicine, and will progressively increase across 24 weeks. Participants will be encouraged to actively cycle at a minimum cadence of ~40-50 rpm, at 40-60% VO2peak for between 10-50 minutes. The intensity of stimulation will be adjusted per leg muscle group based on sensory tolerance with the goal of maintaining pedaling action and target heart rate over the entire session. At each session, we will record the distance traveled, energy expended, power output, resistance, heart rate and rating of perceived exertion (RPE).
  Interventions: Other: FES Cycling Exercise
- Passive Leg Cycling (Placebo Comparator): Passive leg cycling will involve movement of the participant's legs by the cycle ergometer motor without electrical stimulation. The duration of training will follow the same schedule as the FES cycling condition and the same data will be recorded at each session. The passive cycling condition will include the same exposure with the training facility, the exercise equipment (i.e. RT300 cycles), and the research staff (i.e. social contact and attention) as with the FES cycling condition.
  Interventions: Other: Passive Leg Cycling

INTERVENTIONS:
Other: FES Cycling Exercise — FES cycling will use self-adhering surface electrodes (Pals Platinum, Fallbrook, CA) placed over the quadriceps, hamstrings, and gluteal muscle groups to deliver stimulation to the leg muscles.
  Arms: FES Cycling Exercise
Other: Passive Leg Cycling — Passive leg cycling will not involve electrical stimulation
  Arms: Passive Leg Cycling

SUMMARY:
Mobility impairment is one of the most common, poorly managed, and life altering consequences of MS. Current therapies for managing MS do not prevent the long-term accumulation of mobility impairment, highlighting the need for alternative strategies that prevent or slow progressive mobility disability. The proposed trial will test the efficacy and lasting effects of functional electrical stimulation (FES) cycling as an exercise-based rehabilitation strategy for managing mobility impairment and associated consequences in MS.

DETAILED DESCRIPTION:
The study is an assessor-blinded RCT for examining the efficacy and lasting effects of 24 weeks of supervised FES cycling exercise compared to passive leg cycling on mobility and secondary outcomes in people with MS with mobility impairment. Participants who meet the eligibility criteria will undergo the informed consent process and baseline assessment. Participants will then be randomized to either the FES or passive leg cycling program. Following baseline assessment, participants will complete a 24-week leg cycling program, with a mid-point assessment at 12 weeks. At 24 weeks, participants will undergo a post-intervention assessment. Following a 12-week follow-up period, participants will undergo a final assessment. Each participant will be involved in the study for approximately 10 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple sclerosis
* relapse free in the past 30 days
* stable course of disease-modifying therapies over the past 6 months
* ability to communicate in English
* willing to come to the University of Ottawa to complete testing and training sessions
* EDSS score 5.0 - 7.0
* asymptomatic based on a physical activity pre-participation screening tool

Exclusion Criteria:

* presence of any contraindication to FES including epilepsy, a pacemaker, implanted defibrillator, unstable fracture, or pregnancy
* diagnosis of other neurological condition(s)
* participation in FES cycling exercise or other mobility-based exercise rehabilitation program within the past 6 months
* current use of dalfampridine within the past month

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Change in Walking Speed | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Walking speed will be assessed using the timed 25-foot walk (T25FW) test. Participants will walk as quickly and safely as possible across a 25-foot distance (2 trials; average reported in m/s).

SECONDARY OUTCOMES:
Change in Walking Endurance | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Walking endurance will be assessed using the 2-minute walk (2MW) test. Participants will walk as fast and as far as possible in an accessible hallway (1 trial, distance traveled recorded in meters).
Change in Agility | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Agility will be assessed using the Timed Up-and-Go (TUG) test. Participants will rise from a chair, walk 3 meters, turn around, walk back to the chair and return to a seated position (2 trials, time recorded in seconds for both trials)
Change in Patient-rated Mobility Impairment | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Patient-rated impact of MS on walking will be captured using the Multiple Sclerosis Walking Scale-12 (MSWS-12). The MSWS-12 is a 12-item questionnaire that assesses the impact of MS on daily functioning with scores ranging from 0 to 100, where higher scores indicate greater walking impairment.
Change in Cognitive Performance: Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) battery | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  The Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) battery involves three cognitive tasks: the oral version of the Symbol Digit Modalities Test (SDMT), the California Verbal Learning Test II (CVLT-II), and the revised Brief Visualspatial Memory Test (BVMT-R). The SDMT is a timed thinking task that involves associating numbers with symbols. Participants will be asked to provide as many correct numbers as possible in 90 seconds. The CVLT-II is a test of verbal memory and involves recalling a list of words read aloud by an examiner. The participant will be read a list of 16 words and asked to recall as many words as possible. The BVMT is a test of visual memory which involves recalling and manually drawing a series of 6 abstract designs as accurately as possible. The SDMT is performed once, while there are five trials of the CVLT-II and three trials of the BVMT in the BICAMS battery. Higher scores on all three tests indicate better cognitive function.
Change in Cognitive Performance: Paced Auditory Serial Addition Test (PASAT) | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  The Paced Auditory Serial Addition Test (PASAT) involves single numerical digits being presented to a participant every 3 seconds. The participant must add each new digit to the one immediately preceding it. There are 61 numbers presented in total and the total number of correct responses is recorded. Higher scores indicate better cognitive function.
Change in Fatigue Impact | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Fatigue impact will be assessed using the Modified Fatigue Impact Scale (MFIS). The MFIS is a 21-item questionnaire with three subscales (physical, cognitive, and psychosocial), that assess the impact of fatigue on daily functioning over the past 4 weeks. Total MFIS scores are calculated by summing responses for all 21 items, with higher scores indicating greater impact of fatigue. Subscales are calculated based on a subset of items. Scores range from 0-36, 0-40, and 0-8 for physical, cognitive, and psychosocial subscales, respectively, with higher scores indicating greater fatigue.
Change in Fatigue Severity | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Fatigue severity will be assessed by the Fatigue Severity Scale (FSS). The FSS is a nine-item questionnaire that assesses perceived fatigue over the past 7 days. Total FSS scores are calculated as a mean of the nine items. Scores on the FSS range from 1-7, where higher scores indicate more severe fatigue.
Change in Pain | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Pain will be assessed using the McGill Pain Questionnaire (MPQ). The MPQ is a 15-item questionnaire which assesses levels of pain experienced by the participants during a 4-week period. The overall score is calculated by summing responses from each item and can range from 0-45, where higher scores indicate greater severity of pain.
Change in Symptoms of Anxiety and Depression | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Symptoms of anxiety and depression will be assessed using the 14-item Hospital Anxiety and Depression Scale (HADS). The HADS has two subscales (i.e., anxiety and depression) which each contain 7-items, of which a subset are reserve-scored, and then summed into total scores that range from 0-21. Higher scores on each subscale indicate more frequent symptoms of anxiety and depression.
Change in Health-related Quality of Life | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Health-related quality of life will be assessed using the 29-item Multiple Sclerosis Impact Scale (MSIS-29). The MSIS-29 is a measure of physical and psychological health-related QOL. The physical subscale contains 20 items and the psychological subscale contains nine items. Scores from the physical and psychological subscales are computed to range from 0-100, with higher scores indicating a greater physical and psychological impact of MS on daily activities.
Change in Activities of Daily Living | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Participation in activities of daily living will be assessed using the abbreviated Late-Life Function and Disability Instrument (LLFDI). The LLDFI contains 15-items within three subscales: basic lower extremity function, advanced lower extremity function, and upper extremity function. Each subscale contains 5-items and scores range from 5-25. A composite score is generated by summing all three subscale scores, and ranges from 15-75, with higher scores indicating fewer functional limitations.

OTHER OUTCOMES:
Change in Cardiorespiratory Fitness | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Cardiorespiratory fitness will be assessed as peak oxygen consumption based on an incremental exercise test on a recumbent stepper.
Change in Muscular Fitness | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Muscular fitness will be assessed bilaterally as peak torque of the knee extensors/flexors and ankle dorsiflexors/plantarflexors using a Biodex System 4 dynamometer. Peak torque will be obtained by having the participant perform three maximal isometric contractions with each muscle group for 5 seconds, with a 15-second rest between each attempt.
Change in Body Composition | Baseline and 24 weeks
  Body composition will be assessed using dual-energy X-ray absorptiometry (DXA). Data will include percent body fat, fat mass, lean mass, bone mineral density, and bone mineral content.
Change in Optical Coherence Tomography Measures | Baseline, 12 weeks (mid-point), 24 weeks (immediately post intervention), and 36 weeks (12 weeks follow-up)
  Optical coherence tomography (OCT) will be used to capture retinal nerve fibre layer thicknesses.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Pilutti, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards T, Motl RW, Pilutti LA. Cardiorespiratory demand of acute voluntary cycling with functional electrical stimulation in individuals with multiple sclerosis with severe mobility impairment. Appl Physiol Nutr Metab. 2018 Jan;43(1):71-76. doi: 10.1139/apnm-2017-0397. Epub 2017 Sep 7. PMID 28881147
- [Background] Pilutti LA, Motl RW, Edwards TA, Wilund KR. Rationale and design of a randomized controlled clinical trial of functional electrical stimulation cycling in persons with severe multiple sclerosis. Contemp Clin Trials Commun. 2016 May 15;3:147-152. doi: 10.1016/j.conctc.2016.05.005. eCollection 2016 Aug 15. PMID 29736463
- [Background] Edwards T, Motl RW, Sebastiao E, Pilutti LA. Pilot randomized controlled trial of functional electrical stimulation cycling exercise in people with multiple sclerosis with mobility disability. Mult Scler Relat Disord. 2018 Nov;26:103-111. doi: 10.1016/j.msard.2018.08.020. Epub 2018 Sep 8. PMID 30243234